CLINICAL TRIAL: NCT05663203
Title: A Web-Based Dyadic Intervention to Manage Psychoneurological Symptoms for Patients With Colorectal Cancer and Their Caregivers
Brief Title: A Web-Based Dyadic Intervention for Colorectal Cancer
Acronym: CRCweb
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Oncology Nursing Society (Other)
Responsible Party: Principal Investigator, Yufen Lin, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004750; EU5733-22 (Other: Emory University Hospital/Winship Cancer Institute); 2022RE03 (Other Grant/Funding Number: Oncology Nursing Foundation)
Record Dates: First submitted 2022-12-14; First posted 2022-12-23 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (CRCWeb intervention) (Experimental): Patients and caregivers attend a CRCweb intervention over 8 weeks. Patients and caregivers complete interviews and surveys throughout the trial.
  Interventions: Other: Internet-Based Intervention; Other: Interview; Other: Survey Administration; Other: Electronic Health Record Review

INTERVENTIONS:
Other: Internet-Based Intervention — Attend CRCWeb intervention
Other: Interview — Complete interview
Other: Survey Administration — Complete survey
Other: Electronic Health Record Review — Medical records are reviewed

SUMMARY:
This clinical trial studies how well a web-based dyadic intervention works to manage psychoneurological symptoms for patients with colorectal cancer and their caregivers. Patients with colorectal cancer receiving chemotherapy experience severe and distressing psychoneurological symptoms that include fatigue, depression, sleep disturbance, pain, and cognitive dysfunction. When these co-occurring symptoms are undertreated, they negatively affect functional status, survival rates, and quality of life of patients as well as decrease health outcomes of their family caregiver. A critical need exists to develop an effective and novel intervention that focuses on patients with colorectal cancer receiving chemotherapy and their caregivers. A web-based dyadic intervention holds great promise to reduce psychoneurological symptoms burden and improve quality of life for patients with colorectal cancer receiving chemotherapy and advance intervention development and implementation in cancer supportive care and health equity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a web-based dyadic intervention for patients with colorectal cancer receiving chemotherapy and their caregivers (CRCweb).

Ia. Determine tailored contents by identifying needs and supports for a web-based dyadic intervention using interviews with patient-caregiver dyads (n=8); Ib. Develop a prototype of a web-based dyadic intervention program (CRCweb); Ic. Test the usability (e.g., design, navigation, structure, language) of CRCweb prototype using interviews with 4 dyads (in Aim Ia).

II. Evaluate the feasibility and acceptability of CRCweb for patients with colorectal cancer receiving chemotherapy and their caregivers in 20 dyads in a pilot clinical trial.

III. Evaluate the preliminary effects of CRCweb on the primary outcome (i.e., attrition, adherence, acceptability, fatigue, depression, sleep disturbance, pain, and cognitive dysfunction) and secondary outcomes (i.e., quality of life) for patients with colorectal cancer receiving chemotherapy and their caregivers in 20 dyads in a pilot clinical trial.

OUTLINE:

Patients and caregivers attend a CRCweb intervention over 8 weeks. Patients and caregivers complete interviews and surveys throughout the trial.

ELIGIBILITY:
INCLUSION CRITERIA

Patients:

* Age >= 18 years
* Diagnosed with colorectal cancer
* Life expectancy > 12 months
* Receiving active chemotherapy
* Self-reported at least two psychoneurological symptoms (based on the symptom measures' cutoff scores)
* Identified primary caregiver (i.e., family members or significant others identified by the patients as their primary source of emotional and physical support)
* Access to the Internet
* Fluent in English

Caregivers:

* Age >= 18 years
* Primary caregiver
* Access to the Internet
* Fluent in English

EXCLUSION CRITERIA

Patients:

• Karnofsky Performance Scale < 50

Caregivers:

• Have severe diseases (e.g., cancer, heart disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Attrition Rate | Up to week 8
  Collect attendance records from each dyad before and after modules. The intervention will be considered to be high attrition if > 80% dyads remain enrolled. Feasibility of study participation will be assessed by calculating retention rates, identifying reasons for refusal and assessing completeness of the data.
Adherence Rate | Up to week 8
  It is determined by high adherence if dyads complete > 80% of the intervention protocol
Acceptability Rate | Up to week 8
  A survey will be created for this study to assess participants' perceptions of acceptability of the study procedures (> 80% of participants reporting intervention is considered as high acceptability). Participants' perceptions of acceptability of the study procedures and of the intervention itself will be evaluated by calculating descriptive statistics to summarize responses to the post-intervention surveys as well as post-intervention interviews using content analysis.
Multidimensional Fatigue Inventory | Up to week 8
  Fatigue will be measured using the Multidimensional Fatigue Inventory (MFI). The MFI is a 20-item self-reported instrument that includes five dimensions of fatigue: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. Each dimension includes four items on a 1-5 scale. The total score, ranging from 20 to 100 (higher scores indicating more severe fatigue) is calculated as the sum of the five dimensions. The MFI has well established validity and reliability.
Patient Health Questionnaire | Up to week 8
  Depression will be measured using the eight-item Patient Health Questionnaire (PHQ-8), a well-established valid and reliable self-administered diagnostic measure for depressive disorders in clinical studies. The PHQ-8 asks the number of days in the past 2 weeks the respondent has experienced a variety of depressive symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day); the sum of each item is the total score (0 to 24). Patients with a cutoff score of more than 10, clinically significant depression, will be referred to a clinical psychiatrist for further assistance.
Pittsburgh Sleep Quality Index | Up to week 8
  Sleep disturbance will be assessed by the Pittsburgh Sleep Quality Index (PSQI). Its validity and reliability have been established in various populations, including patients with cancer. The PSQI consists of 19 items assessing sleep disturbances in seven dimensions (i.e., subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction). Each dimension scores from 0 (no difficulty) to 3 (severe difficulty), and the sum of these dimension scores is the global sleep quality (0 to 21). Higher scores indicate more difficulty in sleeping.
Brief Pain Inventory | Up to week 8
  Pain will be assessed by the Brief Pain Inventory (BPI). Participants will rate the intensity of the pain (i.e., now, average, worst) using 0 (none) to 10 (excruciating) numeric rating scales (NRS). In addition, they will provide information on the length of time they are in pain, how often their pain occurs, locations of their pain, quality of the pain, pain's level of interference with function, and their level of pain relief and satisfaction with pain treatment.
Attentional Function Index | Up to week 8
  Attentional Function Index (AFI) consists of 16 items designed to measure cognitive dysfunction. A higher total mean score on a 0 to 10 NRS indicates a greater capacity to direct attention. Total scores are grouped into categories of attentional function (i.e., <5.0 low function, 5.0 to 7.5 moderate function, >7.5 high function). In addition, the AFI has three subscales (i.e., effective action, attentional lapses, and interpersonal effectiveness). The AFI has well established reliability and validity.)

SECONDARY OUTCOMES:
Short Form Health Survey | Up to week 8
  The 12-Item Short Form Health Survey (SF-12) consists of 12 questions about physical and mental health as well as overall health status. The individual items on the SF-12 are evaluated and the instrument is scored into two components that measure physical component score and mental component score. These scores can range from 0 to 100. Higher physical component scores and mental component scores indicate a better quality of life. The SF-12 has well established validity and reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Yufen Lin, PhD, RN, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Lin Y, Porter LS, Chee W, Alese OB, Curseen KA, Higgins MK, Northouse L, Xiao C. A Web-Based Dyadic Intervention to Manage Psychoneurological Symptoms for Patients With Colorectal Cancer and Their Caregivers: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2023 Jun 28;12:e48499. doi: 10.2196/48499. PMID 37379055